CLINICAL TRIAL: NCT00308971
Title: Tocopherols and Alpha Lipoic Acid Treatment Chronic Kidney Disease (TALAT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Alp Ikizler, MD, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 051000
Record Dates: First submitted 2006-03-28; First posted 2006-03-30 (Estimated); Last update posted 2009-07-09 (Estimated); Status verified 2009-07

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Gamma Rays; YY1 Transcription Factor; Tocopherols; Vitamin E; Thioctic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Alpha, gamma, beta, and delta (mixed) tocopherols; Drug: alpha lipoic acid
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Alpha, gamma, beta, and delta (mixed) tocopherols — approximately 666 IU daily (1 pill) for 4 months
  Other Names: Vitamin E
  Arms: 1
Drug: alpha lipoic acid — 600 mg daily (2 pills 300 mg each) for 4 months
  Arms: 1
Drug: placebo — placebo for alpha, gamma, beta, and delta (mixed) tocopherols; 1 pill daily for 4 months
  Arms: 2
Drug: placebo — placebo for alpha lipoic acid; 2 pills daily for 4 months
  Arms: 2

SUMMARY:
Oxidative stress and acute phase inflammation are now recognized to be highly prevalent in both the chronic kidney disease (CKD; pre-dialysis) and end stage renal disease (ESRD; on hemodialysis) populations, and several lines of evidence point to their contribution in the development of atherosclerosis. Biomarkers of the inflammatory state such as C-reactive protein (CRP) and interleukin-6 are robust predictors of cardiovascular events and death in these two populations. The uremic state is characterized by retention of oxidized solutes including reactive aldehyde groups and oxidized thiol groups. It has recently been demonstrated that initiation of maintenance hemodialysis does not improve biomarkers of oxidative stress or inflammation, suggesting that dialysis alone is inadequate to control the atherosclerotic uremic metabolic state. In this study we hypothesize that administration of antioxidant therapy will decrease biomarkers of acute phase inflammation and oxidative stress in patients with Stage III and IV CKD.

ELIGIBILITY:
Inclusion criteria:

1. Patients with Stage III-IV chronic kidney disease measured by MDRD formula.
2. age > 18 or < 75 years.
3. Life expectancy greater than one year.
4. Ability to understand and provide informed consent for participation in the study

Exclusion criteria:

1. AIDS (HIV seropositivity is not an exclusion criteria)
2. Active hepatitis C or B
3. Active gout
4. Other active inflammatory diseases.
5. Active malignancy excluding basal or squamous cell carcinoma of the skin.
6. Gastrointestinal dysfunction requiring parental nutrition.
7. History of functional kidney transplant < 6 months prior to study entry.
8. Anticipated live donor kidney transplant over study duration.
9. Prisoners, patients will significant mental illness, pregnant women, and other vulnerable populations.
10. Patients taking Vitamin E supplements > 60 IU/day, vitamin C> 500mg/day over the past 30days.
11. Patients taking anti-inflammatory medication except aspirin < 325mg/day over the past 30 days.
12. Patient taking any prednisone therapy.
13. More than two hospitalizations within the last 90 days or one hospitalization within the last 30 days.
14. On experimental drug protocols.
15. Hypersensitivity to organic nitrates, isosorbide, or nitroglycerin.
16. Hypersensitivity to vitamin E or alpha lipoic acid.
17. Pregnant women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2006-03; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
A statistically significant decrease in F2-isoprostanes, a specific oxidative stress marker | 4 months

SECONDARY OUTCOMES:
A significant change in biomarkers of acute inflammation and oxidative stress from serum | 4 months
A significant change in brachial artery vasodilatation measured by brachial impedence plethysmography | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Himmelfarb, MD, Principal Investigator — MaineHealth; Alp Ikizler, MD, Principal Investigator — Vanderbilt University
Locations (2):
- United States (2):
  - Maine Medical Center, Portland, Maine
  - Vanderbilt University Medical Center, Nashville, Tennessee